CLINICAL TRIAL: NCT00421369
Title: Augmentation of the Antidepressant Action of Sertraline With Triiodothyronine (T3)and Reboxetine: Clinical Efficacy, Adverse Effects and Predictors of Response.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. rena Cooper, HADASSAH MEDICAL ORGANIZATION
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: t3rbx-HMO-CTIL
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2007-01

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Antidepressants; Triiodothyronine (T3); Thyroid Function; Augmentation; Thyroid pathway genes
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sertraline; Triiodothyronine; Reboxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sertraline
Drug: triiodothyronine (T3)
Drug: reboxetine

SUMMARY:
In this project we aim to further refine indications for the use of the thyroid hormone - T3 for patients suffering from depression. We aim to identify a sub-group of patients who are more likely to respond to T3 and establish the time in the treatment course when T3 should be added. The results of this project could have significant, direct clinical implications.

DETAILED DESCRIPTION:
The lifetime risk for major depressive disorder (MDD) is 15% in the general population. Current treatment approaches emphasize the achievement of remission. Remission implies virtual absence of depressive symptoms and is associated with better function and a better overall prognosis than response, which is usually defined as a 50% reduction in symptom severity. Sixty percent or more of patients treated optimally with antidepressants remain un-remitted and will need additional treatment. A potentially effective but under-exploited strategy to augment antidepressant effects is concurrent administration of the thyroid hormone, triiodothyronine (T3). We previously demonstrated the clinical efficacy and safety of T3 administered concurrently with the SSRI, sertraline, in the context of a randomized, double-blind placebo-controlled trial. Although all the patients were euthyroid, remission rates were significantly higher in the sertraline plus T3 group and were associated with significantly lower baseline T3 values and a significant decrease in serum thyroid stimulating hormone (TSH) values during the course of treatment.

The study aims to:

* Delineate a sub-population of depressed patients treated with sertraline, who are more likely to respond to T3 augmentation on the basis of thyroid function and genetic variation in thyroid pathway genes.
* Investigate the appropriate timing for the addition of T3.
* Assess the efficacy of reboxetine, a specific noradrenaline reuptake inhibitor, as a further supplement to the treatment of un-remitted patients. The results of this study could have a significant, direct clinical impact on the pharmacological treatment of MDD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Major Depressive Episode (MDE) in the context MDD according to DSM-IV criteria, without psychotic features.
2. Hamilton Depression Scale (21 items, HAM-D) total >16 with item 1 (depressed mood) >2.
3. Age 18-70 years.
4. Male or female.
5. Competent and willing to give written informed consent.

Exclusion Criteria:

1. Clinical hyper- or hypothyroidism or any other thyroid illness.
2. Neurological or other medical illness that may impact upon the study or limit prescription of the study medications.
3. Significant suicidal risk [HAM-D item 3 (suicide) >2].
4. Comorbidity with any Psychotic Disorder, Bipolar Disorder, Post Traumatic Stress Disorder (PTSD), Eating Disorder.
5. Lifetime history of substance or alcohol dependence or of abuse in the preceding 12 months.
6. Treatment with the antidepressant, sertraline, in current episode.
7. More then one antidepressant trial or any augmentation treatment during current episode.
8. Length of current episode >12 months
9. Female subjects pregnant or lactating or not using adequate contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-09; Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
treatment outcome defined categorically as Remission: A Hamilton Depression Scale (HAM-D) less or equal to 6.

SECONDARY OUTCOMES:
RESPONSE: Based on Hamilton Depression Scale (HAM-D)reduction of >50% from baseline to endpoint..
REMISSION: Based on the other rating scales applied in this project.
RESPONSE: Based on the other rating scales applied in this project.

CONTACTS AND LOCATIONS:
Overall Officials: Rena Cooper-Kazaz, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel